CLINICAL TRIAL: NCT03806621
Title: A Post-Approval Study of the RotablatorTM Rotational Atherectomy System in China
Brief Title: Rota China Registry
Status: Completed | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: BSC International Medical Trading (Shanghai) Co., Ltd. (Other)
Responsible Party: Principal Investigator, Shao-Ping Nie, Professor of Medicine, Director, Center for Coronary Artery Disease, Division of Cardiology, Beijing Anzhen Hospital
Other Study IDs: 2017033
Record Dates: First submitted 2018-12-12; First posted 2019-01-16 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; percutaneous coronary intervention; rotational atherectomy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atherectomy, Coronary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rotational Atherectomy
  Interventions: Procedure: Rotational Atherectomy

INTERVENTIONS:
Procedure: Rotational Atherectomy — Patients with severe calcified lesions will receive rotational atherectomy during index PCI

SUMMARY:
Rotational atherectomy (RA) facilitates percutaneous coronary intervention for complex de novo lesions with severe calcification. Some observational studies and a small randomized trial indicated that a strategy of routine RA did not conferred reduction in restenosis or MACE, but these studies are limited by missing follow-up, insufficient power to compare outcomes, and confounding factors in the RA group (long lesion length, etc.). With recent developments in medical therapy, advances in design and delivery of drug-eluting stents (DES), and advances in noninvasive and intravascular coronary imaging, the use of RA in current real-world practice remains to be well determined. We aimed to compile real-world clinical outcomes data for the RotablatorTM Rotational Atherectomy System in routine clinical practice in China.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Subject who is clinically indicated for PCI/stenting
* Written informed consent
* Subject is willing to comply with all protocol-required follow-up evaluation
* Subject must meet one of following angiographic/procedural inclusion criteria:

  * Target lesion is moderately to severely calcified by visual estimate
  * Unsuccessful balloon dilatation of the target lesion
  * Unsuccessful passage of device(s) (microcatheter, balloon, or stent) across the target lesion

Exclusion Criteria:

* Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute MI within 2 weeks
* Subject has any of the following angiographic findings:

  * Thrombus present in the target vessel (by visual estimate)
  * Significant dissection present in the target vessel (NHLBI types C-F)
  * Lesion angulation > 60°(by visual estimate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This national, multi-center, prospective, observational study will enroll at least 1000 subjects in about 18 to 20 sites in China. All subjects who are candidates for PCI, signed the informed consent form and eligible to receive the treatment using RotablatorTM Rotational Atherectomy System will be evaluated for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 980 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-12-27 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular event (MACE) (primary safety endpoint) | 30 days
  The composite of any ischemia-driven target lesion revascularization (TLR), myocardial infarction (MI), or cardiac death. Periprocedural myocardial infarction, defined as in patients with normal baseline CK-MB, the peak CK-MB measured within 48 hours of the procedure rises to ≥ 10 x the local laboratory ULN, or to ≥ 5 x ULN with new pathologic Q-waves in ≥ 2 contiguous leads or new persistent LBBB (according to SCAI definition. J Am Coll Cardiol 2013;62:1563-70)
Procedural success rate (primary efficacy endpoint) | Peri-procedural
  A mean lesion diameter stenosis <30% in 2 near-orthogonal projections with TIMI 3 flow, as visually assessed by the physician, without the occurrence of in-hospital MI, target vessel revascularization (TVR), or cardiac death

SECONDARY OUTCOMES:
TLR rate | At 30 days and 12 months post-index procedure
Target lesion failure (TLF) rate | At 30 days and 12 months post-index procedure
TVR rate | At 30 days and 12 months post-index procedure
Target vessel failure (TVF) rate | At 30 days and 12 months post-index procedure
MI rate | At 30 days and 12 months post-index procedure
Cardiac death rate | At 30 days and 12 months post-index procedure
Non-cardiac death rate | At 30 days and 12 months post-index procedure
All-cause death rate | At 30 days and 12 months post-index procedure
Cardiac death or MI rate | At 30 days and 12 months post-index procedure
All-cause death or MI rate | At 30 days and 12 months post-index procedure
All-cause death, MI, or TVR rate | At 30 days and 12 months post-index procedure
Stent thrombosis (ST) rate | At 30 days and 12 months post-index procedure
Subgroup analyses of MACE | At 30 days and 12 months post-index procedure
  1. Age (< 65 years vs. ≥ 65 years), 2. Female, 3. Hypertension, 4. Diabetes, 5. CKD, 6. Left ventricular ejection fraction (≤ 50% vs. > 50%), 7. LM lesion, 8. Long lesion, 9. CTO, 10. Bifurcation lesion, 11. Speed of rotation, 12. Maximal burr size, 13. IVUS or OCT use

OTHER OUTCOMES:
Rate of arterial perforation (rotational atherectomy related or non-related) | Peri-procedural
Rate of abrupt coronary occlusion (including dissection and thrombosis) | Peri-procedural
Rate of significant coronary dissection (NHLBI types C-F) | Peri-procedural
Rate of consistent no reflow | Peri-procedural

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangdong Academy of Medical Science, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing First hospital, Nanjing Medical University, Nanjing, Jiangsu
  - First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xijing Hospital, the Fourth Military Medical University, Xi'an, Shaanxi
  - Qilu Hospital (Qingdao), Shandong University, Jinan, Shandong
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Fourth Central Hospital, Tianjin, Tianjin Municipality
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Wang X, Zhang H, Bai X, Zhang L, Li C, Mao X, Chen J, Luo J, Zhao Y, Zhou B, You B, Zhang Y, Ma L, Du Z, Chen Y, Sun F, Qiu C, Shen Z, Wen S, Mintz GS, Ye F, Nie S; China Rota Elite Group. Practices and outcomes of rotational atherectomy in China: The Rota China registry. Catheter Cardiovasc Interv. 2024 Oct;104(4):664-675. doi: 10.1002/ccd.31211. Epub 2024 Sep 3. PMID 39223992